CLINICAL TRIAL: NCT00961766
Title: Phase 1: A Single-Center, Randomized, Blinded, Placebo-Controlled, Single-Administration, Sequential-Cohort, Dose-Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of BG00010 (Neublastin) Administered to Sciatica Participants
Brief Title: Evaluate the Safety, Tolerability and Pharmacokinetics of BG00010 (Neublastin) Administered to Sciatica Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103NS101
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BG00010 (Neublastin) (Experimental): Participants may be randomized to escalating doses of BG00010 or matching placebo
  Interventions: Drug: BG00010 (Neublastin)
- Placebo (Placebo Comparator): Participants may be randomized to escalating doses of BG00010 or matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG00010 (Neublastin) — Single dose, weight-based IV administration
  Arms: BG00010 (Neublastin)
Drug: Placebo — Single dose IV matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the safety/tolerability profile, systemic PK behavior, and immunogenicity of single IV and SC administrations of BG00010 to sciatica participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of unilateral sciatica, determined by the Investigator. Sciatica symptoms must be present for 6 or more weeks prior to the Screening Visit.
* Must have a body mass index (BMI) between 18 kg/m2 and 32 kg/m2.
* Must rate their pain at >40 mm on the 100 mm Visual Analog Scale (VAS) of the Short-Form McGill Pain Questionnaire (SF-MPQ)at the Screening and Baseline Visits.

Key Exclusion Criteria:

* History of malignancy or clinically significant (as determined by the Investigator) allergies, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (not related to sciatica), dermatologic, rheumatic/joint, psychiatric, renal, and/or other major disease.
* History of signs or symptoms of peripheral neuropathy, other than symptoms of sciatica.
* History of severe allergic or anaphylactic drug-related reactions. NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing Adverse Events (AEs) | Up to 56 days post dosing
Change in Likert numerical pain rating scale | Up to 56 days post dosing
Change in Quantitative Sensory Test (QST) | Up to 28 days post dosing
  QST; Vibratory, Cool Thermal,
Change in Intra Epidermal Nerve Fiber Density (IENFD) | Up to 28 days post dosing
Maximum observed serum concentration (Cmax) | Up to 5 days post dosing
Area under the serum concentration curve (AUC) | Up to 5 days post dosing
Terminal half-life (t1/2) | Up to 5 days post dosing
Total body clearance (CL) | Up to 5 days post dosing
Steady state volume of distribution (Vss) | Up to 5 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Rolan PE, O'Neill G, Versage E, Rana J, Tang Y, Galluppi G, Aycardi E. First-In-Human, Double-Blind, Placebo-Controlled, Randomized, Dose-Escalation Study of BG00010, a Glial Cell Line-Derived Neurotrophic Factor Family Member, in Subjects with Unilateral Sciatica. PLoS One. 2015 May 11;10(5):e0125034. doi: 10.1371/journal.pone.0125034. eCollection 2015. PMID 25962165